CLINICAL TRIAL: NCT07228260
Title: Help Texts Grief Intervention for Bereaved College Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Arizona (Other); Help Texts (Industry)
Responsible Party: Principal Investigator, Ted Robles, PhD, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-25-0709
Record Dates: First submitted 2025-09-23; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Bereavement
Keywords: bereavement; digital intervention; text-based intervention; college students

STUDY DESIGN:
Intervention Model Description: The treatment group will receive the Help Texts intervention at baseline, whereas the waitlist control group will receive treatment as usual (list of resources for grief) at baseline. At 6 months, the waitlist control group will receive the Help Texts intervention as well.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist Control with Treatment as Usual (Other): At study enrollment, participants receive treatment as usual--a list of resources relevant to grief.
  At 6 months following study enrollment, participants will receive a 12-month subscription to Help Texts, a text-based intervention that delivers two texts per week providing bereavement psychoeducation, validation, and coping strategies.
  Interventions: Behavioral: list of resources for grief; Behavioral: text-based intervention for grief
- Treatment (Active Comparator): At study enrollment, participants will receive a 12-month subscription to Help Texts, a text- based intervention that delivers two texts per week providing bereavement psychoeducation, validation, and coping strategies.
  Interventions: Behavioral: text-based intervention for grief

INTERVENTIONS:
Behavioral: list of resources for grief — Participants will receive treatment as usual, consisting of a list of resources for coping with grief both on-campus and off-campus
  Arms: Waitlist Control with Treatment as Usual
Behavioral: text-based intervention for grief — Help Texts delivers texts twice a week over a period of 12-months to provide psychoeducation, validation, and coping strategies relevant to bereavement. The The texts offer some customization in specifying the name of the participant and their deceased loved one, as well as providing texts relevant to the participants' cause of bereavement and relationship to their deceased loved one.
  Other Names: Help Texts

SUMMARY:
The proposed study aims to evaluate the effectiveness of Help Texts, a weekly text-based program, among bereaved students at UCLA. Specifically, the study will evaluate whether Help Texts reduces grief severity and symptoms of depression, and whether it improves academic functioning (e.g., graduation, grades, student enrollment retention).

The investigators hypothesize that bereaved UCLA students who receive a 12-month Help Texts weekly digital text intervention will have reduced grief severity and depressive symptoms and increased academic functioning compared to bereaved UCLA students in a waitlist control condition receiving treatment as usual (i.e., list of resources for grief).

Participants will complete surveys at four timepoints: baseline and 3 months, 6 months, and 12 months following enrollment. They will be randomly assigned to either the treatment condition (receive 12-month Help Texts subscription at enrollment) or the waitlist control condition (receive list of resources for grief at enrollment, and receive 12-month Help Texts subscription at 6 months following enrollment). The Help Texts program involves texts offering psychoeducation related to grief and coping strategies, delivered twice weekly.

DETAILED DESCRIPTION:
Grief and loss are common occurrences among students on college campuses but are inadequately addressed and associated with a number of negative outcomes. A mixed methods study of grieving students on a large campus found that 60% of those surveyed within a 3-year period at UCLA reported experiencing the loss of a loved one, but only 8% reported using campus resources to aid them during their grief, and only 38% sought resources off-campus (e.g., therapy, support groups, psychiatry). Numerous barriers to accessing grief support resources have been identified, including not knowing about them or perceiving them to be inadequate. Moreover, over one-third of participants interviewed in the study noted stigma associated with help-seeking. Despite a high prevalence of experiences of grief among students, resource utilization for supporting bereavement remains low.

Help Texts offers text message-based grief support, overcoming the barriers of access and stigma by providing up to a year of private, evidence-based grief support developed by clinical psychologists. Help Texts is an established company (specifically, a Public Benefit Corporation) and is currently in use. It was founded in 2018 and comprises a fully remote, 7-person team with over 100+ additional Expert Contributors providing expertise on different types of loss (e.g., the loss of a sibling, child, parent, partner; loss to cancer, dementia, suicide, COVID-19, etc); and the unique risks associated with being a caregiver, veteran, or member of the LGBTQIA2S+ or Black, Indigenous, and People of Color (BIPOC) communities. Help Texts is delivering support in 57 countries, in all 50 states in the U.S., and in 27 languages.

Help Texts provides twice-weekly, one-way texts offering basic grief education by normalizing and validating the grief experience and then offering tips for coping within various themes around grief. Preliminary evidence suggests that bereaved users of HelpTexts have found it supportive; 95% of all users rated their satisfaction with HelpTexts as a 4 or 5 out of 5 and found the text messages helpful. The proposed study is a randomized control trial that aims to evaluate the effectiveness of Help Texts to grieving students at UCLA in reducing grief severity and symptoms of depression, preventing prolonged grief and major depressive disorder, and in improving quality of life and occupational functioning (e.g., graduation, grades, student enrollment retention).

ELIGIBILITY:
Inclusion Criteria:

* Enrolled UCLA student
* At least 18 years old
* Experienced death of a close person in the past 12 months
* Able to read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Prolonged Grief Disorder-Revised (PG-13-R) | 0 months, 3 months, 6 months, 12 months following enrollment
  PG-13-R measures symptoms of Prolonged Grief Disorder (PGD) mapping onto the Diagnostic and Statistical Manual's conceptualization of clinical grief. The measure assesses symptoms such as yearning for the deceased close person, avoiding reminders of their death, and feelings of loneliness in relation to the death. Each item is rated from 1 (Not at all) to 5 (Overwhelmingly). Total scores range from 10 to 50, with higher scores representing more severe prolonged grief.
Patient Health Questionnaire (PHQ-3) | 0 months, 3 months, 6 months, 12 months following enrollment
  The PHQ-3 measures symptoms of depression over the last 2 weeks, including loss of interest in things, feeling down or hopeless, and feeling tired. Each item is rated from 0 (Not at all) to 3 (Nearly every day). Total scores range from 0 to 9, with higher scores representing more severe symptoms of depression.

SECONDARY OUTCOMES:
Academic Functioning - GPA | 0 months, 3 months, 6 months, 12 months following enrollment
  Participants' current overall GPA will be measured. From highest to lowest, the GPA options will be the following: A+, A, A-, B+, B, B-, C+, C, C-, D+ or below, with A+ representing the highest possible current overall GPA.
Academic Functioning - Negative Impacts to Academic Performance | 0 months, 3 months, 6 months, 12 months following enrollment
  The investigators will assess the number of days that participants felt that emotional or mental difficulties hurt their academic performance. Participants can select the following options: None (0), 1-2 days (1), 3-5 days (2), 6 or more days (3), with scores ranging from 0 to 3. Higher scores indicate more days that participants felt their academic performance was hurt by their emotional or mental difficulties.
Academic Functioning - Class Enrollment Status | 0 months, 3 months, 6 months, 12 months following enrollment
  Participants will indicate whether or not they are currently registered for classes at UCLA. They will respond Yes (1) or No (0), with a higher score indicating that they are currently registered for classes.
Academic Functioning - Dropped Course | 0 months, 3 months, 6 months, 12 months following enrollment
  Another academic outcome measured will be whether or not participants dropped a course in the past quarter. This will be dichotomously scored as Yes (1) or No (0), with a higher score indicating endorsement of having dropped a course in the past quarter.

OTHER OUTCOMES:
Generalized Anxiety Disorder-7 (GAD-7) | 0 months, 3 months, 6 months, 12 months following enrollment
  The GAD-7 will assess symptoms of generalized anxiety over the past 2 weeks consistent with the Diagnostic and Statistical Manual's conceptualization of generalized anxiety. It will assess symptoms such as being unable to control worrying and having difficulty relaxing. Items will be scored from 0 (Not at all) to 3 (Nearly every day). Total scores will range from 0 to 21, with higher scores indicating more severe symptoms of generalized anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Franz Hall, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Our data will be securely managed by members of our research team and will not be shared with members outside of our research team. Findings from our research will be summarized and shared such that participants are not individually identifiable. Should other collaborators desire to access our data, they will need to be aligned with the goals of our research and added and approved to our IRB protocol.

REFERENCES:
- [Result] Levesque DA, Lunardini MM, Adams SN, Payne EL, Neumann BG. Grief Coach: Feasibility and acceptability of a text message program for bereavement support among grievers in the United Kingdom. Death Stud. 2025;49(4):391-402. doi: 10.1080/07481187.2024.2334080. Epub 2024 Apr 4. PMID 38573792
- [Result] Chang M, Panda S, Tajrian M, Kim WI, Dunkel Schetter C, Robles TF. Bereavement, resource utilization, and collective grieving since the COVID pandemic: Mixed-methods study of university students and staff. 2024.
- [Result] Varga MA, Lanier B, Biber D, Stewart B. Holistic Grief Effects, Mental Health, and Counseling Support in Bereaved College Students. College Student Affairs Journal. 2021;39(1):1-13. doi: 10.1353/csj.2021.0000.
- [Result] Sirrine EH, Kliner O, Gollery TJ. College Student Experiences of Grief and Loss Amid the COVID-19 Global Pandemic. Omega (Westport). 2023 Aug;87(3):745-764. doi: 10.1177/00302228211027461. Epub 2021 Jun 23. PMID 34162233
- [Result] Jones S, Martini M. Sense of self, depression and adaption to grief, in emerging adults who suffered parental loss. Current Psychology. 2023;42(7):5212-25. doi: 10.1007/s12144-021-01843-z.